CLINICAL TRIAL: NCT02810951
Title: A Phase I/II Study of FCX-007 (Genetically-Modified Autologous Human Dermal Fibroblasts) for Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Brief Title: A Study of FCX-007 for Recessive Dystrophic Epidermolysis Bullosa (RDEB)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Subjects were all in Long-Term Follow Up and were transferred to the ongoing EB-002 study
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FI-EB-001; FD-R-6113-01 (Other Grant/Funding Number: Office of Orphan Products Development)
Record Dates: First submitted 2016-06-13; First posted 2016-06-23 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Epidermolysis Bullosa Dystrophica, Recessive
Keywords: RDEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FCX-007 (Experimental): In Phase I, a target of three adult subjects will be enrolled into Group A and a target of three adult subjects will be enrolled into Group B.
  In Phase II the study will target enrolling subjects (aged seven (7 years or older) to each arm, but will allow a disproportionate distribution of subjects between Group A and Group B to equal approximately 6 total subjects.
  All subjects will receive FCX-007 into one or more paired target wounds as well as to intact skin at least one time during the study with a possible second administration pending laboratory results.
  One wound in each target wound pair will be used as control for efficacy and safety evaluations.
  Interventions: Genetic: FCX-007

INTERVENTIONS:
Genetic: FCX-007 — FCX-007 is a genetically modified cell product obtained from the subject's own skin cells (Autologous fibroblasts). The cells are expanded and genetically modified to produce functional COL7. FCX-007 cell suspension is injected intradermally.
  Other Names: Genetically-Modified Autologous Human Dermal Fibroblasts

SUMMARY:
The purpose of this study is to evaluate the safety of FCX-007, evaluate Type VII collagen (COL7) expression and the presence of anchoring fibrils and to analyze wound healing as a result of FCX-007 administration in subjects with recessive dystrophic epidermolysis bullosa (RDEB). Funding Source- FDA OOPD

DETAILED DESCRIPTION:
RDEB is a rare skin and connective tissue disease characterized clinically by skin fragility with easy blistering, erosion and scarring of skin and mucous membranes, and caused by the deficiency of the protein type VII collagen (COL7). The objective of this study is evaluate the safety of FCX-007 intradermal injections in RDEB subjects. Additionally, the trial will evaluate COL7 expression, the presence of anchoring fibrils, as well evidence of wound healing.

Approximately twelve subjects are expected to enroll in the Phase I/II trial. Phase I will enroll approximately six adult subjects. Phase II will enroll approximately six subjects both adults and pediatric (aged seven (7) years or older). All subjects will receive FCX-007 to one or more paired target RDEB wounds. Proof of mechanism will be monitored through digital photography of target wounds and assays conducted on biopsies taken from intact skin sites where FCX-007 is administered.

ELIGIBILITY:
Key Inclusion Criteria:

1. Age

   1. Phase I: Eighteen (18) years or older.
   2. Phase II: Seven (7) years or older.
2. Diagnosis of recessive dystrophic epidermolysis bullosa (RDEB)

Key Exclusion Criteria:

1. Medical instability limiting ability to travel to the investigative center.
2. Active infection with HIV, hepatitis B or hepatitis C or evidence of other systemic infection
3. Current evidence of metastatic squamous cell carcinoma at the site to be injected
4. Clinically significant abnormal laboratory result or other significant clinical abnormalities
5. Receipt of a chemical or biological study product for the specific treatment of RDEB in the past six months

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All subjects will receive FCX-007 intradermal injections into a treated wound in a target pair and will have no FCX-007 injections into the other control wound in the target pair.
Period: Overall Study
Arm/Group | All Study Participants
Started | 6
FCX-007 Injection | 6
No FCX-007 Injection | 6
Completed | 5
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- FCX-007: In Phase I, a target of three adult subjects will be enrolled into Group A and a target of three adult subjects will be enrolled into Group B.
  In Phase II the study will target enrolling subjects (aged seven (7) or older) to each arm, but will allow a disproportionate distribution of subjects between Group A and Group B to equal approximately 6 total subjects.
  All subjects will receive FCX-007 into intact skin as well as to one or more paired target wounds at least one time during the study with a possible second administration pending laboratory results.
  One wound in each target wound pair will be used as control for efficacy and safety evaluations. FCX-007 administered wounds will be compared within paired target wounds to untreated wounds.
  FCX-007: FCX-007 is a genetically modified cell product obtained from the subject's own skin cells (Autologous fibroblasts). The cells are expanded and genetically modified to produce functional collagen VII. FCX-007 cell suspension is injected intradermally.
Arm/Group | FCX-007
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 28.4 [9.1 to 38.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Open target wounds [Number; unit: number of wounds] | 10

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of subjects with adverse events.
Time Frame: 52 weeks post treatment
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Who Received FCX-007 Injections: All subjects who received FCX-007 injections in at least one target wound.
Arm/Group | Subjects Who Received FCX-007 Injections
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Complete Wound Closure
Description: Percentage of target wounds achieving complete wound closure (greater than 90%) at all post-baseline visits
Time Frame: Through Week 52
Population: Number analyzed represents observed wounds/participants only
Measure: Number; unit: percentage of target wounds
Units Other Than Participants: target wounds
Groups:
- Treated Wounds: FCX-007 is a genetically modified cell product obtained from the subject's own skin cells (Autologous fibroblasts). The cells are expanded and genetically modified to produce functional collagen 7 (COL7). FCX-007 cell suspension is injected intradermally.
- Untreated Wounds: No FCX-007 injected
Arm/Group | Treated Wounds | Untreated Wounds
Number analyzed (Participants) | 6 | 6
Number analyzed (target wounds) | 10 | 10
percentage of target wounds
  Complete closure at Week 4 | 40.0 | 0
  Complete closure at Week 12: number analyzed (target wounds) | 10 | 9
  Complete closure at Week 12 | 80.0 | 0
  Complete closure at Week 25: number analyzed (Participants) | 2 | 2
  Complete closure at Week 25: number analyzed (target wounds) | 4 | 4
  Complete closure at Week 25 | 75.0 | 0
  Complete closure at Week 52: number analyzed (Participants) | 4 | 4
  Complete closure at Week 52: number analyzed (target wounds) | 6 | 6
  Complete closure at Week 52 | 50.0 | 16.7

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Adverse events were reported on the whole participant level and not segmented to treated or control wounds
Arm/Group | FCX-007
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCX-007 (N=6)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCX-007 (N=6)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site discolouration (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed for proof of mechanism analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02810951/Prot_SAP_000.pdf